CLINICAL TRIAL: NCT02016560
Title: An Open Label, Multicenter Study, Evaluating the Safety and Imaging Characteristics of 18F-AV-1451 in Cognitively Healthy Volunteers, Subjects With Mild Cognitive Impairment, and Subjects With Alzheimer's Disease
Brief Title: Analysis of 18F-AV-1451 PET Imaging in Cognitively Healthy, MCI, and AD Subjects
Acronym: MCI
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Avid Radiopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Diagnostic
Other Study IDs: 18F-AV-1451-A05
Record Dates: First submitted 2013-12-16; First posted 2013-12-20 (Estimated); Results first posted 2020-08-24 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — florbetapir; 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole

STUDY DESIGN:
Intervention Model Description: All subjects in both the exploratory and confirmatory phases of the study, receive both florbetapir and florbetapir scans, regardless of subgroup assignment.
Who Masked: Outcomes Assessor
Masking Description: Applies only to confirmatory phase: the independent readers are blinded to all clinical information.
Oversight: Data Monitoring Committee: No

ARMS (4):
- Exploratory Cognitively Healthy Subjects (Experimental): Subjects will receive an IV injection, 370 megabecquerel (MBq) (10 millicurie [mCi]), single dose of florbetapir F 18 at baseline. Subjects will receive an IV injection, 370 MBq (10 mCi), single dose of flortaucipir at baseline.
  Interventions: Drug: florbetapir F 18; Drug: Flortaucipir F18; Procedure: Brain PET Scan
- Exploratory MCI Subjects (Experimental): Subjects will receive an IV injection, 370 MBq (10 mCi), single dose of florbetapir F 18 at baseline. Subjects will receive an IV injection, 370 MBq (10 mCi), single dose of flortaucipir at baseline, 9 months and 18 months.
  Interventions: Drug: florbetapir F 18; Drug: Flortaucipir F18; Procedure: Brain PET Scan
- Exploratory AD Subjects (Experimental): Subjects will receive an IV injection, 370 MBq (10 mCi), single dose of florbetapir F 18 at baseline. Subjects will receive an IV injection, 370 MBq (10 mCi), single dose of flortaucipir at baseline, 9 months and 18 months.
  Interventions: Drug: florbetapir F 18; Drug: Flortaucipir F18; Procedure: Brain PET Scan
- Confirmatory Subjects (Experimental): Subjects will receive an IV injection, 370 MBq (10 mCi), single dose of florbetapir F 18 and flortaucipir at baseline.
  Interventions: Drug: florbetapir F 18; Drug: Flortaucipir F18; Procedure: Brain PET Scan

INTERVENTIONS:
Drug: florbetapir F 18
  Other Names: Amyvid; 18F-AV-45
Drug: Flortaucipir F18
  Other Names: T807; 18F-AV-1451
Procedure: Brain PET Scan — positron emission tomography (PET) scan of the brain

SUMMARY:
A Phase 2/3 cross-sectional and longitudinal observational study evaluating imaging characteristics of flortaucipir in control subjects and patients with clinically defined MCI and AD dementia (AD).

DETAILED DESCRIPTION:
This study was conducted in 2 phases: a Phase 2 Exploratory Phase and a Phase 3 Confirmatory Phase. An overarching goal of the Exploratory Phase of this protocol was to further investigate the pattern of flortaucipir PET imaging across the disease course, in cognitively healthy subjects through patients with cognitive decline. To accomplish this goal, the protocol investigated flortaucipir results in younger and older cognitively healthy normal volunteers and patients with clinical diagnoses for cognitive complaints, ranging from MCI to mild and moderate AD dementia. Additionally, the Exploratory Phase of this protocol investigated relationships between flortaucipir PET signal and cognitive decline over the 18-month study period.

The second, Confirmatory Phase of the study was designed to provide independent validation of the relationships observed in the exploratory analyses of the first phase. In particular, the goal of the second phase was to confirm the relationship between flortaucipir uptake in the brain as measured by PET signals at baseline and the subsequent rate of cognitive decline observed over the 18-month longitudinal follow up.

ELIGIBILITY:
Inclusion Criteria:

Exploratory Cognitively Healthy Subjects

* ≥ 20 to ≤ 40 years of age OR ≥ 50 years of age
* Mini-mental state examination (MMSE) ≥ 29
* No significant history of cognitive impairment

Exploratory MCI Subjects

* ≥ 50 years of age
* MMSE ≥ 24
* Have MCI consistent with National Institute on Aging-Alzheimer's Association (NIA-AA) working group's diagnostic guidelines for AD
* Have a study partner that can report on subject's activities of daily living

Exploratory AD Subjects

* ≥ 50 years of age
* MMSE > 10
* Have possible or probable AD based on the NIA-AA working group's diagnostic guidelines for AD
* Have a study partner that can report on subject's activities of daily living

Confirmatory Subjects

* ≥ 50 years of age
* MMSE ≥ 20 and ≤ 27
* Cognitively impaired subjects with either MCI or dementia with a suspected neurodegenerative cause
* Have a study partner that can report on subject's activities of daily living

Exclusion Criteria:

* Current clinically significant psychiatric disease
* Evidence of structural brain abnormalities
* History of moderate or severe traumatic brain injury
* Current clinically significant cardiovascular disease or ECG abnormalities, or additional risk factors for Torsades de Pointes
* Current clinically significant infectious disease, endocrine or metabolic disease, pulmonary, renal or hepatic impairment, or cancer
* History of alcohol or substance abuse or dependence
* Females of childbearing potential who are not surgically sterile, not refraining from sexual activity or not using reliable methods of contraception
* Have received or participated in a trial with investigational medications in the past 30 days
* Have had a non-study related radiopharmaceutical imaging or treatment procedure within 7 days prior to the study imaging session.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 383 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2017-07-28 (Actual); Study Completion 2017-07-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (27):
- United States (27):
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Four Peaks Neurology, Scottsdale, Arizona
  - Mayo Clinic, Scottsdale, Arizona
  - Banner Sun Health Research Institute, Sun City, Arizona
  - UC Irvine, Irvine, California
  - Hoag Memorial, Newport Beach, California
  - Norther California PET Imaging Center, Sacramento, California
  - UC Davis, Sacramento, California
  - UC San Francisco, San Francisco, California
  - Neurological Research Institute, Santa Monica, California
  - Molecular NeuroImaging, New Haven, Connecticut
  - Quantum Laboratories, Deerfield Beach, Florida
  - 21st Century Oncology, Fort Myers, Florida
  - Sandlake Imaging, Orlando, Florida
  - Meridien Research, St. Petersburg, Florida
  - USF Health Byrd Alzheimer's Center, Tampa, Florida
  - Independent Imaging, West Palm Beach, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston University, Boston, Massachusetts
  - Alzheimer's Disease Center, Quincy, Massachusetts
  - Center for Clinical Imaging Research, St Louis, Missouri
  - Las Vegas Radiology, Las Vegas, Nevada
  - Center for Brain Health - NYU Langone Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Butler Hospital, Providence, Rhode Island

REFERENCES:
- [Derived] Lu M, Pontecorvo MJ, Devous MD Sr, Arora AK, Galante N, McGeehan A, Devadanam C, Salloway SP, Doraiswamy PM, Curtis C, Truocchio SP, Flitter M, Locascio T, Devine M, Zimmer JA, Fleisher AS, Mintun MA; AVID Collaborators. Aggregated Tau Measured by Visual Interpretation of Flortaucipir Positron Emission Tomography and the Associated Risk of Clinical Progression of Mild Cognitive Impairment and Alzheimer Disease: Results From 2 Phase III Clinical Trials. JAMA Neurol. 2021 Apr 1;78(4):445-453. doi: 10.1001/jamaneurol.2020.5505. PMID 33587110

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Exploratory cohort subjects were enrolled starting in Dec 2013. Confirmatory cohort subjects were enrolled Dec 2014-July 2017. Exploratory cohort subjects were not eligible for the confirmatory phase.
Pre-assignment Details: To ensure a distribution of disease severity in the confirmatory phase, a target was set to recruit at least one-third of the enrolled subjects with dementia
Groups:
- Exploratory Young Cognitively Healthy Subjects: Male or female subjects ≥20 to ≤40 years of age with mini-mental status exam (MMSE) score ≥29
- Exploratory Older Cognitively Healthy Subjects: Male or female subjects ≥50 years of age with MMSE Score ≥29
- Exploratory MCI Subjects: Subjects with mild cognitive impairment consistent with National Institute of Aging (NIA)-Alzheimer's Association working group's diagnostic guidelines for AD (Albert et al. 2011) and MMSE Score ≥24
- Exploratory AD Subjects: Subjects with possible or probable AD dementia based on the NIA-Alzheimer's Association working group's diagnostic guidelines for AD (McKhann et al. 2011) and MMSE Score >10
- Confirmatory Subjects MCI: Clinically diagnosed mild cognitive impairment with a suspected neurodegenerative cause with an MMSE score ≥20 and ≤27
- Confirmatory Subjects AD: Clinically diagnosed dementia with a suspected neurodegenerative cause with an MMSE score ≥20 and ≤27
Period: Exploratory Phase
Arm/Group | Exploratory Young Cognitively Healthy Subjects | Exploratory Older Cognitively Healthy Subjects | Exploratory MCI Subjects | Exploratory AD Subjects | Confirmatory Subjects MCI | Confirmatory Subjects AD
Started | 16 | 58 | 98 | 51 | 0 | 0
Completed | 16 | 54 | 62 | 35 | 0 | 0
Not Completed | 0 | 4 | 36 | 16 | 0 | 0
Period: Confirmatory Phase
Arm/Group | Exploratory Young Cognitively Healthy Subjects | Exploratory Older Cognitively Healthy Subjects | Exploratory MCI Subjects | Exploratory AD Subjects | Confirmatory Subjects MCI | Confirmatory Subjects AD
Started | 0 | 0 | 0 | 0 | 98 | 62
Completed | 0 | 0 | 0 | 0 | 76 | 35
Not Completed | 0 | 0 | 0 | 0 | 22 | 27

BASELINE CHARACTERISTICS:
Groups:
- Exploratory Young Cognitively Healthy Subjects: Male or female subjects ≥20 to ≤40 years of age with MMSE ≥29
- Exploratory Older Cognitively Healthy Subjects: Male or female subjects ≥50 years of age with MMSE ≥29
- Exploratory MCI Subjects: Subjects with mild cognitive impairment consistent with National Institute of Aging (NIA)-Alzheimer's Association working group's diagnostic guidelines for AD (Albert et al. 2011) and MMSE ≥24
- Exploratory AD Subjects: Subjects with possible or probable AD dementia based on the NIA-Alzheimer's Association working group's diagnostic guidelines for AD (McKhann et al. 2011) and MMSE >10
- Total: Total of all reporting groups
Arm/Group | Exploratory Young Cognitively Healthy Subjects | Exploratory Older Cognitively Healthy Subjects | Exploratory MCI Subjects | Exploratory AD Subjects | Confirmatory Subjects MCI | Confirmatory Subjects AD | Total
Number analyzed (Participants) | 16 | 58 | 98 | 51 | 98 | 62 | 383
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age, Continuous for Exploratory Cohort only
  years
    number analyzed (Participants) | 16 | 58 | 98 | 51 | 0 | 0 | 223
    (all) | 28.9 (4.88) | 68.5 (10.29) | 70.8 (9.3) | 73.9 (9.01) |  |  | 67.9 (14.36)
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age, Continuous for Confirmatory Cohort only
  years
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 98 | 62 | 160
    (all) |  |  |  |  | 72.5 (9.69) | 73.6 (9.53) | 72.9 (9.61)
Sex: Female, Male [Count of Participants; unit: Participants] — Exploratory Cohort - Sex: Female, Male
  Participants
    Female | 7 | 26 | 49 | 28 | 44 | 30 | 184
    Male | 9 | 32 | 49 | 23 | 54 | 32 | 199
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 4 | 0 | 5 | 4 | 15
  Not Hispanic or Latino | 15 | 57 | 94 | 51 | 93 | 58 | 368
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 1 | 1 | 0 | 1 | 1 | 5
  Black or African American | 3 | 9 | 7 | 2 | 3 | 0 | 24
  White | 11 | 47 | 89 | 47 | 94 | 61 | 349
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Other | 1 | 1 | 1 | 1 | 0 | 0 | 4
Clinical Dementia Rating - Sum of Boxes (CDR-SB) [Mean (Standard Deviation); unit: units on a scale] — The CDR scale (Berg 1988) examines 6 cognitive functioning domains individually on a scale of 0 to 3. CDR Sum of Boxes is generated by summing the total score across domains. Scores range from 0 to 18, with higher scores indicating higher levels of cognitive impairment. Population: Recorded at baseline only for confirmatory phase subjects
  units on a scale
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 98 | 61 | 159
    (all) |  |  |  |  | 2.8 (1.73) | 4.3 (1.69) | 3.4 (1.88)

OUTCOME MEASURES:

1. Primary Outcome: Confirmatory Phase: Relationship Between Neocortical Flortaucipir Uptake and the Subsequent Rate of Cognitive Decline
Description: Confirm the relationship between neocortical flortaucipir uptake and the subsequent rate of cognitive decline at longitudinal follow up that was observed in the Exploratory Phase of the study. Patients were assigned to groups by majority classification of the flortaucipir positron emission tomography (PET) scan by five independent imaging physicians. Clinically meaningful cognitive and functional deterioration was defined as a 1 point or greater worsening on clinical dementia rating - sum of boxes (CDR-SB) score over the follow-up period.
Time Frame: between baseline and 18 months
Population: Subjects from the confirmatory phase with valid flortaucipir visual read and 9 or 18 month clinical follow-up.
Measure: Count of Participants; unit: Participants
Groups:
- Predicted to Progress: Subjects with an Advanced AD Scan Pattern (τAD++). In either hemisphere, increased neocortical activity in the parietal/precuneus region(s), or frontal region(s) with increased uptake in the PLT, parietal, or occipital region(s).
- Not Predicted to Progress: Subjects with a Moderate AD Scan Pattern (τAD+) or Not AD Scan Pattern (τAD-). Moderate scans were defined as in either hemisphere, increased neocortical activity limited to the posterolateral temporal (PLT) or occipital region(s). Not AD scans were defined as no increased neocortical activity, or increased neocortical activity isolated to the mesial temporal, anterolateral temporal, and/or frontal regions.
Arm/Group | Predicted to Progress | Not Predicted to Progress
Number analyzed (Participants) | 63 | 68
Participants
  Clinically meaningful progression | 36 | 31
  Did Not Progress | 27 | 37
Statistical Analysis 1: Comparison: Predicted to Progress vs Not Predicted to Progress; The specific hypothesis tested was that the hazard of progressing to the clinically meaningful event (defined as CDR-SB value change of at least 1 within 18 months) will be significantly greater for subjects with flortaucipir scans rated by majority interpretation as predicted to progress (Advanced AD scan pattern), as compared to subjects with scans rated as not predicted to progress (Moderate or Not AD scan pattern); Test type: Other; p = 0.067, Cox proportional hazards — A p-value of <0.05 was the a priori threshold for statistical significance; The Cox proportional hazard model was adjusted for baseline age, American National Adult Reading Test (ANART) score, and baseline CDR-SB score; Cox Proportional Hazard = 1.581, 95% CI 2-sided [0.968 to 2.581]

2. Primary Outcome: Exploratory Phase: Cross-sectional Flortaucipir Imaging Results
Description: Flortaucipir standardized uptake value ratio (SUVr). A value of 1 signifies no flortaucipir activity above background, values greater than 1 signify increasing flortaucipir activity in the brain.
Time Frame: baseline scan
Population: Analysis included all subjects who received an injection of flortaucipir, had valid quantifiable flortaucipir imaging data available, and valid quantifiable florbetapir PET data.
Measure: Least Squares Mean (Standard Error); unit: standardized uptake value ratio (SUVr)
Arm/Group | Exploratory AD Subjects | Exploratory MCI Subjects | Exploratory Older Cognitively Healthy Subjects | Exploratory Young Cognitively Healthy Subjects
Number analyzed (Participants) | 48 | 97 | 57 | 16
standardized uptake value ratio (SUVr)
  Aβ+ SUVr: number analyzed (Participants) | 32 | 47 | 5 | 0
  Aβ+ SUVr | 1.53 (0.037) | 1.26 (0.030) | 1.08 (0.093) |
  Aβ- SUVr: number analyzed (Participants) | 16 | 50 | 52 | 16
  Aβ- SUVr | 1.03 (0.051) | 0.99 (0.029) | 0.98 (0.029) | 1.01 (0.039)
Statistical Analysis 1: Comparison: Exploratory AD Subjects vs Exploratory Older Cognitively Healthy Subjects; ANCOVA model comparing the mean SUVr between AD and Older Cognitively Healthy within amyloid positive group; Test type: Other; p < 0.0001, ANCOVA — No adjustment for multiple comparisons. No a priori threshold was set; Adjusted for age
Statistical Analysis 2: Comparison: Exploratory MCI Subjects vs Exploratory Older Cognitively Healthy Subjects; ANCOVA model comparing the mean SUVr between MCI and Older Cognitively Healthy within the amyloid positive group; Test type: Other; p = 0.0622, ANCOVA — No adjustment for multiple comparisons. No a priori threshold was set; Adjusted for age
Statistical Analysis 3: Comparison: Exploratory AD Subjects vs Exploratory MCI Subjects; ANCOVA model comparing the mean SUVr between AD and MCI within the amyloid positive group; Test type: Other; p < 0.0001, ANCOVA — No adjustment for multiple comparisons. No a priori threshold was set; Adjusted for age

3. Primary Outcome: Exploratory Phase: Longitudinal Change in Tau Deposition Over Time, by Amyloid Status
Description: Assess the rate of change of tau deposition as measured by flortaucipir uptake (SUVr) over time. Change = 18 months SUVr - baseline SUVr.
Time Frame: baseline and 18 months
Population: Analysis of flortaucipir SUVr Change Over Time by Amyloid Status, Exploratory Phase Efficacy Population (AD and MCI subjects only)
Measure: Least Squares Mean (Standard Error); unit: standardized uptake value ratio (SUVr)
Groups:
- Exploratory AB+ (Amyloid Beta Positive): Exploratory MCI or AD subjects with a positive florbetapir PET scan for amyloid
- Exploratory AB- (Amyloid Beta Negative): Exploratory MCI or AD subjects with a negative florbetapir PET scan for amyloid
Arm/Group | Exploratory AB+ (Amyloid Beta Positive) | Exploratory AB- (Amyloid Beta Negative)
Number analyzed (Participants) | 55 | 90
standardized uptake value ratio (SUVr) | 0.052359 (0.008536) | 0.000655 (0.002394)
Statistical Analysis 1: Comparison: Exploratory AB+ (Amyloid Beta Positive); SUVr change from baseline as dependent variable, baseline SUVr, age, and visit as independent variables, using an unstructured covariance structure for amyloid positive subjects only; Test type: Equivalence — Test of whether the least squares mean change is significantly different than zero; p < 0.0001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Exploratory AB- (Amyloid Beta Negative); SUVr change from baseline as dependent variable, baseline SUVr, age, and visit as independent variables, using an unstructured covariance structure for amyloid negative subjects only; Test type: Equivalence — Test of whether the least squares mean change is significantly different than zero; p = 0.7851, Mixed Models Analysis

4. Secondary Outcome: Confirmatory Phase: Diagnostic Performance of Flortaucipir Visual Read
Description: This analysis used dichotomized CDR-SB change as a truth standard (1 point or more worsening = true positive vs. less than 1 point worsening = true negative) to assess the diagnostic performance of baseline Advanced AD tau status (τAD++) as determined by flortaucipir scan interpretation. Sensitivity and Specificity were calculated for each of the 5 independent imaging readers. Sensitivity is the percentage of true positive cases correctly identified by an Advanced AD pattern scan. Specificity is the percentage of true negative cases correctly identified by scans that were not classified as Advanced AD pattern.
Time Frame: baseline and 18 months
Population: All confirmatory phase subjects who completed 18 months of follow-up for the cognitive endpoint were read by each reader
Measure: Number (95% Confidence Interval); unit: percentage of cases correctly identified
Groups:
- Independent Readers: Scans were interpreted by 5 imaging physicians, blind to clinical data, after training by an Avid expert.
Arm/Group | Independent Readers
Number analyzed (Participants) | 110
percentage of cases correctly identified
  Reader 1 Sensitivity: number analyzed (Participants) | 52
  Reader 1 Sensitivity | 59.6 [46.1 to 71.8]
  Reader 1 Specificity: number analyzed (Participants) | 58
  Reader 1 Specificity | 65.5 [52.7 to 76.4]
  Reader 2 Sensitivity: number analyzed (Participants) | 52
  Reader 2 Sensitivity | 53.8 [40.5 to 66.7]
  Reader 2 Specificity: number analyzed (Participants) | 58
  Reader 2 Specificity | 65.5 [52.7 to 76.4]
  Reader 3 Sensitivity: number analyzed (Participants) | 52
  Reader 3 Sensitivity | 55.8 [42.3 to 68.4]
  Reader 3 Specificity: number analyzed (Participants) | 58
  Reader 3 Specificity | 65.5 [52.7 to 76.4]
  Reader 4 Sensitivity: number analyzed (Participants) | 52
  Reader 4 Sensitivity | 59.6 [46.1 to 71.8]
  Reader 4 Specificity: number analyzed (Participants) | 58
  Reader 4 Specificity | 65.5 [52.7 to 76.4]
  Reader 5 Sensitivity: number analyzed (Participants) | 52
  Reader 5 Sensitivity | 50.0 [36.9 to 63.1]
  Reader 5 Specificity: number analyzed (Participants) | 58
  Reader 5 Specificity | 65.5 [52.7 to 76.4]
Statistical Analysis 1: Comparison: Independent Readers; Test type: Other; The hypothesis tested was that, of the 5 independent imaging physicians, at least 3 will have the lower bounds of 2-sided 95% confidence intervals ≥50%, for both sensitivity and specificity

5. Secondary Outcome: Exploratory Phase: Correlation Between Flortaucipir SUVr and Age
Description: as for outcome 2
Time Frame: baseline scan
Population: Exploratory Young and Old healthy control subjects with a valid flortaucipir PET scan
Measure: Mean (Standard Deviation); unit: standardized uptake value ratio (SUVr)
Groups:
- Exploratory Older Cognitively Healthy Subjects 50-59: Male or female subjects 50-59 years of age with MMSE ≥29
- Exploratory Older Cognitively Healthy Subjects 60-69: Male or female subjects 60-69 years of age with MMSE ≥29
- Exploratory Older Cognitively Healthy Subjects 70-79: Male or female subjects 70-79 years of age with MMSE ≥29
- Exploratory Older Cognitively Healthy Subjects >=80: Male or female subjects 80 years of age or older with MMSE ≥29
Arm/Group | Exploratory Young Cognitively Healthy Subjects | Exploratory Older Cognitively Healthy Subjects 50-59 | Exploratory Older Cognitively Healthy Subjects 60-69 | Exploratory Older Cognitively Healthy Subjects 70-79 | Exploratory Older Cognitively Healthy Subjects >=80
Number analyzed (Participants) | 16 | 15 | 15 | 16 | 11
standardized uptake value ratio (SUVr) | 1.0083 (0.03905) | 1.0203 (0.03693) | 1.0110 (0.04149) | 1.0010 (0.02604) | 1.0048 (0.03978)
Statistical Analysis 1: Comparison: Exploratory Young Cognitively Healthy Subjects vs Exploratory Older Cognitively Healthy Subjects 50-59 vs Exploratory Older Cognitively Healthy Subjects 60-69 vs Exploratory Older Cognitively Healthy Subjects 70-79 vs Exploratory Older Cognitively Healthy Subjects >=80; Pearson's correlation coefficient; Test type: Other; p = 0.4361, Pearson; Pearson's correlation coefficient = -0.0925

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected at scan visits, regardless of attribution to study drug. End of study for AE reporting was 48 hours after the last study drug administration. AEs occurring after study drug administration, but outside that window were not recorded, unless considered attributable to either drug.
Groups:
- Exploratory Younger Cognitively Healthy Subjects: Male or female subjects ≥20 to ≤40 years of age with MMSE ≥29
Arm/Group | Exploratory Younger Cognitively Healthy Subjects | Exploratory Older Cognitively Healthy Subjects | Exploratory MCI Subjects | Exploratory AD Subjects | Confirmatory Subjects MCI | Confirmatory Subjects AD
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/58 | 0/98 | 0/51 | 0/98 | 0/62
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/58 | 1/98 | 0/51 | 0/98 | 0/62
Other Adverse Events (participants affected / at risk) | 3/16 | 17/58 | 21/98 | 13/51 | 13/98 | 0/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exploratory Younger Cognitively Healthy Subjects (N=16) | Exploratory Older Cognitively Healthy Subjects (N=58) | Exploratory MCI Subjects (N=98) | Exploratory AD Subjects (N=51) | Confirmatory Subjects MCI (N=98) | Confirmatory Subjects AD (N=62)
angina pectoris (Cardiac disorders) | 0 (0) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Exploratory Younger Cognitively Healthy Subjects (N=16) | Exploratory Older Cognitively Healthy Subjects (N=58) | Exploratory MCI Subjects (N=98) | Exploratory AD Subjects (N=51) | Confirmatory Subjects MCI (N=98) | Confirmatory Subjects AD (N=62)
Angina pectoris (Cardiac disorders) | 0 | 1 | 2 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Injection site pain (General disorders) | 0 | 5 | 8 | 2 | 6 | 0
Injection site extravasation (General disorders) | 0 | 0 | 3 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 2 | 1 | 0 | 0 | 0
Application site irritation (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Application site laceration (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Feeling abnormal (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Therapeutic response unexpected (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Blood pressure increased (Investigations) | 0 | 2 | 2 | 1 | 0 | 0
Blood pressure systolic increased (Investigations) | 0 | 2 | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0
Heart rate increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 3 | 3 | 1 | 4 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 2 | 0
Head discomfort (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 2 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cyanopsia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (4):
  • Study Protocol (2015-08-07): https://cdn.clinicaltrials.gov/large-docs/60/NCT02016560/Prot_000.pdf
  • Statistical Analysis Plan: Confirmatory Phase SAP (2018-01-05): https://cdn.clinicaltrials.gov/large-docs/60/NCT02016560/SAP_001.pdf
  • Statistical Analysis Plan: Confirmatory Phase Addendum SAP (2018-01-05): https://cdn.clinicaltrials.gov/large-docs/60/NCT02016560/SAP_002.pdf
  • Statistical Analysis Plan: Exploratory Phase SAP (2017-11-27): https://cdn.clinicaltrials.gov/large-docs/60/NCT02016560/SAP_003.pdf